CLINICAL TRIAL: NCT04881747
Title: Bioequivalence of Lasmiditan Oral Disintegrating Tablet Compared to Current Immediate-Release Tablet Formulation to Support Treatment of Migraine
Brief Title: A Study to Compare Two Different Formulations of Lasmiditan in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 17016; H8H-MC-LAIA (Other: Eli Lilly and Company)
Record Dates: First submitted 2021-05-10; First posted 2021-05-11 (Actual); Results first posted 2023-03-23 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2021-08

CONDITIONS: Healthy
MeSH Terms: interventions — lasmiditan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 100 milligram (mg) Lasmiditan immediate release (IR) (Reference) (Active Comparator): Participants received 100 mg lasmiditan as IR tablet formulation administered orally.
  Interventions: Drug: Lasmiditan
- 100 mg Lasmiditan oral disintegrating (OD) Without Water (Test) (Experimental): Participants received 100 mg lasmiditan as OD tablet formulation administered orally without water.
  Interventions: Drug: Lasmiditan
- 100 mg Lasmiditan OD With Water (Test) (Experimental): Participants received 100 mg lasmiditan as OD tablet formulation administered orally with water.
  Interventions: Drug: Lasmiditan

INTERVENTIONS:
Drug: Lasmiditan — Administered orally.
  Other Names: LY573144

SUMMARY:
The main purpose of this study is to compare the amount of lasmiditan that gets into the blood stream and how long it takes the body to get rid of it, when given as a oral-disintegrating (OD) tablet compared to immediate-release (IR) tablet formulation. The information about any adverse effects experienced will be collected and the tolerability of lasmiditan when administered as OD tablet will also be evaluated.

Screening is required within 28 days prior to the start of the study. For each participant, the total duration of the clinical trial will be about 5 weeks, including screening.

ELIGIBILITY:
Inclusion Criteria:

* Are overtly healthy as determined by medical evaluation.
* Body mass index (BMI) of 19 to 35 kilograms per meter squared (kg/m²).

Exclusion Criteria:

* Have known allergies to lasmiditan, related compounds, or any components of the formulation of lasmiditan, or a history of significant atopy.
* Have an abnormal blood pressure and/or pulse rate, as determined by the investigator.
* Have clinically significant abnormalities on ECG, as determined by investigator.
* Have a history or presence of cardiovascular, respiratory, renal, gastrointestinal, endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; of constituting a risk when taking the study interventions; or of interfering with the interpretation of data.
* Have used or are intending to use over-the-counter or prescription medication, including dietary supplements, within 14 days prior to dosing and until study discharge (apart from occasional acetaminophen, hormonal contraception, or hormone-replacement therapy).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2021-05-14 (Actual); Primary Completion 2021-07-24 (Actual); Study Completion 2021-07-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Covance Dallas, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Crossover study with three study periods, each participant received immediate release (IR) tablet as reference; oral disintegrating (OD) tablet with water and without water as test doses of 100 milligram (mg) lasmiditan according to their assigned treatment sequence, on Day 1 of each Period. The washout period between dosing in consecutive study periods was approximately 5 days.
Groups:
- Sequence 1: Participants received lasmiditan on day 1 of each treatment period as per the below dosing sequence:
  Period 1: 100 mg lasmiditan IR; Period 2: 100 mg lasmiditan OD without water; and Period 3: 100 mg lasmiditan OD with water.
- Sequence 2: Participants received lasmiditan on day 1 of each treatment period as per the below dosing sequence:
  Period 1: 100 mg lasmiditan IR; Period 2: 100 mg lasmiditan OD with water; and Period 3: 100 mg lasmiditan OD without water.
- Sequence 3: Participants received lasmiditan on day 1 of each treatment period as per the below dosing sequence:
  Period 1: 100 mg lasmiditan OD without water; Period 2: 100 mg lasmiditan OD with water; and Period 3: 100 mg lasmiditan IR.
- Sequence 4: Participants received lasmiditan on day 1 of each treatment period as per the below dosing sequence:
  Period 1: 100 mg lasmiditan OD without water; Period 2: 100 mg lasmiditan IR; and Period 3: 100 mg lasmiditan OD with water.
- Sequence 5: Participants received lasmiditan on day 1 of each treatment period as per the below dosing sequence:
  Period 1: 100 mg lasmiditan OD with water; Period 2: 100 mg lasmiditan IR; and Period 3: 100 mg lasmiditan OD without water.
- Sequence 6: Participants received lasmiditan on day 1 of each treatment period as per the below dosing sequence:
  Period 1: 100 mg lasmiditan OD with water; Period 2: 100 mg lasmiditan OD without water; and Period 3: 100 mg lasmiditan IR.
Period: Period 1
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6
Started | 8 | 8 | 8 | 8 | 8 | 7
Received At Least One Dose of Study Drug | 8 | 8 | 8 | 8 | 8 | 7
Completed | 8 | 8 | 8 | 8 | 8 | 7
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 1 Washout
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6
Started | 8 | 8 | 8 | 8 | 8 | 7
Completed | 8 | 8 | 8 | 8 | 8 | 7
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 2
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6
Started | 8 | 8 | 8 | 8 | 8 | 7
Received At Least One Dose of Study Drug | 8 | 8 | 8 | 8 | 8 | 7
Completed | 8 | 8 | 8 | 8 | 8 | 7
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 2 Washout
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6
Started | 8 | 8 | 8 | 8 | 8 | 7
Completed | 6 | 8 | 8 | 7 | 7 | 7
Not Completed | 2 | 0 | 0 | 1 | 1 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 1 | 0 | 0
Period: Period 3
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6
Started | 6 | 8 | 8 | 7 | 7 | 7
Received At Least One Dose of Study Drug | 6 | 8 | 8 | 7 | 7 | 7
Completed | 6 | 8 | 8 | 7 | 7 | 7
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6 | Total
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 7 | 47
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.6 (13.3) | 35.6 (12.5) | 40.6 (14.3) | 35.8 (12.6) | 43.5 (11.5) | 47.3 (12.5) | 40.4 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 4 | 2 | 3 | 2 | 16
  Male | 6 | 5 | 4 | 6 | 5 | 5 | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 2 | 1 | 2 | 2 | 10
  Not Hispanic or Latino | 7 | 6 | 6 | 7 | 6 | 5 | 37
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 1 | 1 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 5 | 4 | 5 | 4 | 4 | 2 | 24
  White | 3 | 4 | 3 | 3 | 3 | 5 | 21
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 8 | 8 | 8 | 8 | 8 | 7 | 47

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics (PK): Maximum Concentration (Cmax) of Lasmiditan
Description: PK: Cmax of Lasmiditan.
Time Frame: Predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8,12, 24, 48, 72, 96 and 120 hours post-dose
Population: All enrolled participants who received at least one dose of study drug (lasmiditan) and had evaluable pharmacokinetic data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Groups:
- 100 mg Lasmiditan IR (Reference): Participants received 100 mg lasmiditan as IR tablet formulation administered orally.
- 100 mg Lasmiditan OD Without Water (Test): Participants received 100 mg lasmiditan as OD tablet formulation administered orally without water.
Arm/Group | 100 mg Lasmiditan IR (Reference) | 100 mg Lasmiditan OD Without Water (Test) | 100 mg Lasmiditan OD With Water (Test)
Number analyzed (Participants) | 46 | 46 | 44
nanograms per milliliter (ng/mL) | 140 (43) | 123 (42) | 124 (43)
Statistical Analysis 1: Comparison: 100 mg Lasmiditan IR (Reference) vs 100 mg Lasmiditan OD Without Water (Test); Test type: Equivalence — Model: Log(PK) = Treatment + Sequence + Period + Participant(Sequence) + Random Error, where participant within sequence is fitted as a random effect; Ratio of Geometric least squares mean = 0.875, 90% CI 2-sided [0.834 to 0.919]
Statistical Analysis 2: Comparison: 100 mg Lasmiditan IR (Reference) vs 100 mg Lasmiditan OD With Water (Test); Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of Geometric least squares mean = 0.889, 90% CI 2-sided [0.846 to 0.934]

2. Primary Outcome: PK: Area Under the Concentration Versus Time Curve From Time Zero to Infinity (AUC[0-inf]) of Lasmiditan
Description: PK: AUC[0-inf] of Lasmiditan.
Time Frame: Predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8,12, 24, 48, 72, 96 and 120 hours post-dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng*h/ mL)
Arm/Group | 100 mg Lasmiditan IR (Reference) | 100 mg Lasmiditan OD Without Water (Test) | 100 mg Lasmiditan OD With Water (Test)
Number analyzed (Participants) | 46 | 46 | 44
nanogram*hour per milliliter (ng*h/ mL) | 937 (39) | 884 (39) | 881 (39)
Statistical Analysis 1: Comparison: 100 mg Lasmiditan IR (Reference) vs 100 mg Lasmiditan OD Without Water (Test); Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of Geometric least squares mean = 0.944, 90% CI 2-sided [0.914 to 0.976]
Statistical Analysis 2: Comparison: 100 mg Lasmiditan IR (Reference) vs 100 mg Lasmiditan OD With Water (Test); Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of Geometric least squares mean = 0.946, 90% CI 2-sided [0.914 to 0.978]

3. Primary Outcome: PK: Area Under the Plasma Concentration Versus Time Curve From Time Zero to the Last Measured Concentration Value (AUC[0-tlast]) of Lasmiditan
Description: PK: AUC[0-tlast] of Lasmiditan.
Time Frame: Predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8,12, 24, 48, 72, 96 and 120 hours post-dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | 100 mg Lasmiditan IR (Reference) | 100 mg Lasmiditan OD Without Water (Test) | 100 mg Lasmiditan OD With Water (Test)
Number analyzed (Participants) | 46 | 46 | 44
ng*h/mL | 915 (39) | 860 (39) | 860 (39)
Statistical Analysis 1: Comparison: 100 mg Lasmiditan IR (Reference) vs 100 mg Lasmiditan OD Without Water (Test); Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of Geometric least squares mean = 0.941, 90% CI 2-sided [0.910 to 0.972]
Statistical Analysis 2: Comparison: 100 mg Lasmiditan IR (Reference) vs 100 mg Lasmiditan OD With Water (Test); Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of Geometric least squares mean = 0.944, 90% CI 2-sided [0.913 to 0.977]

ADVERSE EVENTS:
Time Frame: Baseline, Up to 49 days
Description: All enrolled participants who received at least one dose of study drug (lasmiditan).
Arm/Group | 100 mg Lasmiditan IR (Reference) | 100 mg Lasmiditan OD Without Water (Test) | 100 mg Lasmiditan OD With Water (Test)
All-Cause Mortality (participants affected / at risk) | 0/47 | 0/46 | 0/44
Serious Adverse Events (participants affected / at risk) | 0/47 | 0/46 | 0/44
Other Adverse Events (participants affected / at risk) | 0/47 | 0/46 | 0/44

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2020-09-08): https://cdn.clinicaltrials.gov/large-docs/47/NCT04881747/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-10): https://cdn.clinicaltrials.gov/large-docs/47/NCT04881747/SAP_001.pdf